CLINICAL TRIAL: NCT06081192
Title: Accuracy and Clinical Outcomes of Titanium-zirconium One-piece Mini Implants Using a Partially-guided Surgery for Maxillary Overdentures: a Pilot Prospective Clinical Study
Brief Title: Partially-guided Protocol for Maxillary Overdentures Retained by Ti-Zr One-piece Mini Implants
Acronym: SMIS-Max
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Goias (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Full Professor, Universidade Federal de Goias
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI07294-2023
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Edentulous Jaw; Implant Complication
Keywords: Dental implant; Overdenture; Edentulous patient; Clinical study; Effectiveness
MeSH Terms: conditions — Jaw, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Single-center, single-group, prospective clinical trial
Masking Description: Not applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-piece titanium-zirconium mini implants (Experimental): Six one-piece titanium-zirconium mini implants (Straumann® Mini Implant System, Institut Straumann AG, Switzerland) in the edentulous maxilla, using a partially-guided insertion protocol.
  Interventions: Procedure: Implant placement surgery

INTERVENTIONS:
Procedure: Implant placement surgery — Placement of six mini implants in the edentulous maxilla using a partially-guided protocol
  Other Names: Dental implant

SUMMARY:
This is a single-center, single-group, prospective clinical trial testing a partially-guided protocol for placement of mini implants overdentures in the edentulous maxilla. Eligible participants will be subjects with an edentulous maxilla, wearing a conventional complete denture. Participants will receive six mini implants (Straumann® Mini Implant System, Institut Straumann AG, Switzerland) for retention of a maxillary overdenture. The six mini implant protocol will be virtually planned for an even distribution of the implants bilaterally, with a minimum of 5 mm distance between contiguous implants. The available lengths of the mini implants are 10, 12, and 14 mm, and the appropriate length will be selected according to the bony anatomical situation. In addition, the distribution and axial position of the mini implants will be planned to achieve the best biomechanical distribution and the most parallel position between implants, perpendicular to the occlusal plane and path of insertion of the prosthesis. The primary outcome will be the accuracy of the implant position using the partially-guided protocol. Assessment of the accuracy of the methods will be based on the measure of the difference between the actual and the planned position of the mini implants, based on the measurement of (1) the global deviations at the coronal and apical regions of the mini implants, (2) the vertical deviation, and (3) the apical angle deviation. Overall impacts of treatment on oral health-related quality of life will be assessed using the Oral Health Impact Profile instrument for edentulous subjects (OHIP-EDENT). Additional outcomes will include implant survival and success rates, incidence of prosthodontic complications and peri-implant measurements.

DETAILED DESCRIPTION:
Design This is a single-center, single-group, prospective clinical trial testing a partially-guided protocol for placement of mini implants overdentures in the edentulous maxilla.

Study setting, trial registration, and funding This clinical trial will be conducted in the clinical setting of the School of Dentistry of the Federal University of Goias, Brazil. The research protocol will be previously submitted for ethical approval by the local Ethical Research Committee and will be registered prospectively at the ClinicalTrial.gov database before initiating patient recruitment.

Participants Eligible participants will be subjects with an edentulous maxilla, wearing a conventional complete denture. They will be selected from the list of patients who received conventional treatment at least six months previously. The possible conditions of the mandibular arch will include fully dentate subjects, partially edentate wearing fixed or removable prostheses, fixed or removable implant-supported dentures, or a shortened dental arch.

During the recruitment phase of the study, they will be informed about the treatment to be provided, details about the clinical trial, and the need for collaboration in the prescribed procedures and post-treatment follow-up visits over a minimum 1-year period. The selected participants will sign an informed consent form to participate in the study.

Inclusion and exclusion criteria We will select participants ≥ 60 years of age, with an edentulous maxillary arch, wearing a complete maxillary denture evaluated as sufficient for surgical planning. At the implant site level, they should present a healed edentulous maxilla (minimum of twelve weeks since the last extraction), minimal ridge dimensions of 5.4 mm (width) by 12 mm (height) in the anterior and premolar maxillary area, allowing the placement of one-piece implants with a 2.4 mm-diameter and minimum length of 10 mm. General health condition should be a physical status ASA1 or ASA2.

Excluded criteria will comprise the inability to perform adequate oral hygiene, incapability to provide written informed consent and compliance to the protocol, and any contraindication for oral surgery such as but not limited to, uncontrolled diabetes, immunosuppression, radiation, chemotherapy, or antiresorptive medication such as bisphosphonates, presence of dental, periodontal or peri-implant disease in the opposing arch, presence of a conventional complete denture in the opposing arch (mandible), presence of an insufficient partial removable denture or implant-overdenture in the opposing arch, which cannot be rendered sufficient by a reline, a heavy smoking habit with > 20 cig/d, reported severe bruxism or clenching habits, clinically present oro-facial pain, depression with a Geriatric Depression Scale above 12, xerostomia with a stimulated salivary flow rate inferior to 0.7 ml/min. At the implant site level, potential participants will be excluded if they present a ridge morphology type IV, defects requiring bone augmentation procedures, or unhealthy soft tissues.

Intervention This prospective clinical trial will be conducted on maxillary edentulous patients recruited for treatment with six mini implants (Straumann® Mini Implant System, Institut Straumann AG, Switzerland) for retention of a maxillary overdenture.

Surgical diagnostic will consist of a preoperative visit with a thorough examination of the patient's medical and dental history, and clinical and radiological assessment. This includes a preliminary OPT-tomography to determine ridge morphology and exclude patients with insufficient ridge dimensions before additional radiographic examinations. In case of a positive preliminary radiographical examination, the radiological analysis will be performed with a Cone Beam Computed Tomography (CBCT) radiograph of the maxillary arch. The existing denture will be marked with gutta-percha or composite spheres in the second premolar, canine and central incisor regions prior to image-taking for the purpose of spatial reference. The existing denture will be subsequently scanned with an intra-oral scanner (TRIOS; 3 Shape), and the STL file will be imported into an implant planning software (coDiagnostiX; Dental Wings GmbH) along with the DICOM files of the CBCT. The six mini implant protocol will be virtually planned for an even distribution of the implants bilaterally, with a minimum of 5 mm distance between contiguous implants. The available lengths of the mini implants are 10, 12, and 14 mm, and the appropriate length will be selected according to the bony anatomical situation. In addition, the distribution and axial position of the mini implants will be planned to achieve the best biomechanical distribution and the most parallel position between implants, perpendicular to the occlusal plane and path of insertion of the prosthesis.

Outcomes

1. Accuracy of implant placement The primary outcome will be the accuracy of the implant position using the partially-guided protocol. Assessment of the accuracy of the methods will be based on the measure of the difference between the actual and the planned position of the mini implants, based on the measurement of (1) the global deviations at the coronal and apical regions of the mini implants, (2) the vertical deviation, and (3) the apical angle deviation. The global deviation is defined as the 3D distance between the coronal/apical centers of the planned and placed implants. The vertical deviation is the distance between the coronal center of the longitudinal axis of the planned implant and a plane parallel through the coronal center of the placed implant. The angle deviation will be measured as the angular divergence between the longitudinal axes of the planned and actual position of the mini implants.

   For image assessment, post-operative CBCT will be performed six weeks after surgery using the same CBCT machine and protocol used for the pre-operative CBCT. The images of the pre- and post-operative CBCTs will be superimposed using the automated surface best fit matching with the iterative closest point algorithm in the treatment evaluation mode of the coDiagnostiX® software. The individual deviations for the six inserted mini implants will be measured (in millimeters) at the limit between the machined and SLA surface of the mini implant, and at the apex between the planned and actual implant positions. The divergence of the implant axis (in degrees) will also be recorded. Six separate superimposing scans of the CBCT image will be obtained for each of the mini implants inserted in each patient, and measurements of deviations and angulations will be done separately.
2. Treatment intercurrencies and complications Any complications associated with the surgical procedures, or deviations from the prescribed protocol due to surgical intercurrences will be recorded. These include failed drilling of the planned implant site, need to raise a flap for adequate positioning of the needle drill, fracture of the bone walls, insufficient insertion torque (< 10 Ncm), early implant failure, and others.
3. Patient-reported outcomes (PROs) Overall impacts of treatment on oral health-related quality of life will be assessed using the Oral Health Impact Profile instrument for edentulous subjects (OHIP-EDENT). This is a shorter version of the 49-item OHIP, and the validated Portuguese translation of the questionnaire will be utilized.

   Denture satisfaction will be evaluated by using the Denture Satisfaction Index (DSI), a 10mm visual analogue scale (VAS)-based questionnaire. This index evaluates ease of cleaning, general satisfaction, speech, comfort, aesthetics, stability, chewing ability, function and the general oral condition.
4. Chewing efficiency Chewing efficiency will be evaluated with a two-color mixing ability test, where participants are given a two-colored chewing gum and are asked to chew the specimen for 20 chewing cycles. The resulting bolus is evaluated visually on a reference scale and opto-electronically using the Variance of Hue (VOH).
5. Maximum voluntary bite force (MBF) The Gnathodynamometer DMD® (Kratos Equipamentos Industriais Ltda., Cotia - SP, Brazil) is utilized. It is a digital force gauge with an 8.6mm thick bite element. MBF is assessed bilaterally between the upper and lower first molar. The participant's task is to bite as hard as possible on the force gauge, but to stop clenching when she/ he starts feeling uncomfortable. The peak force of three recordings carried out on each side will be used for analysis.
6. Implant Survival and Success

   Implant Survival and Success rate will be defined as followed:

   I - Success (optimum health) II - Satisfactory survival III - Compromised survival

   IV - Failure (clinical absolute failure) Any of following:

   Additionally, fractured implants will be considered as failures, except fracture of the implant apex during implant placement.
7. Prosthetic Success and Survival

   During the prosthodontic examination, the implant-supported prostheses will be examined for any complications according to the 2015 ITI Treatment Guide:

   A failure will be defined as an event leading to the loss of the reconstruction and need for the fabrication of a new overdenture.
8. Clinical Peri-implant Measurements At 4 sites per implant (mesial/distal/buccal/oral), the following clinical parameters will be evaluated at baseline and each follow-up visit: Plaque index and bleeding on probing; Pocket probing depth; width of the keratinized tissue around implants.
9. Peri-implant bone height Intra-oral radiographs are exported and four parallel lines are drawn corresponding to the shoulder and the apical end of the implant on. One line each is placed at the shoulder and apical end of the implant and the other two at the defined bone level on the mesial and distal aspect of the implant. Knowing the implant length and using the implant-shoulder as a reference point, bone levels can be calculated through a simple rule of three with NIH Image J V1.44.
10. Implant Stability Primary implant stability will be assessed by measuring the final and peak insertion torques, and the primary and secondary implant stability will be assessed using the Periotest® instrument.

The Periotest® hand piece (Periotest®, Siemens AG, Bensheim, Germany) will be used with the head of the patient stabilized so that the implants were perpendicular to the floor, and the Periotest will be held parallel to the floor. The test point will be in the most gingival region of the Optiloc attachment, and each measurement will be performed 3 times and the average value will be recorded for each implant.

Sample size:

The sample size for this study will include 10 participants. A 20% increase in sample size will be adopted to account for patient dropout during the 1-year follow-up, and with no relevant impact on the study power. Therefore, the final sample will comprise of 12 participants, and 72 units at the implant-level.

Data analysis:

Descriptive statistics and bivariate tests for independent groups will be used to analyze differences between groups, according to the data distribution patterns. Subsequently, a Linear Mixed-Effects Model (LMM) regression will be used to test the effect of independent variables (anatomic and functional features) on the post-surgical accuracy of the implant position. This multi-level approach will be used because of the clustered effect of multiple implants within patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age
* healed dentulous maxillary arch (minimum of twelve weeks since the last extraction)
* wearing a complete maxillary denture evaluated as sufficient for surgical planning
* minimal ridge dimensions of 5.4 mm (width) by 12 mm (height) in the anterior and premolar maxillary area
* bone dimensions allowing the placement of one-piece implants with a 2.4 mm-diameter and minimum length of 10 mm.
* general health condition should be a physical status ASA1 or ASA2.

Exclusion Criteria:

* inability to perform adequate oral hygiene
* incapability to provide written informed consent and compliance to the protocol
* any contraindication for oral surgery such as but not limited to,

  * uncontrolled diabetes
  * immunosuppression
  * radiation or chemotherapy
  * antiresorptive medication such as bisphosphonates
  * presence of dental, periodontal or peri-implant disease in the opposing arch
  * presence of a conventional complete denture in the opposing arch (mandible)
  * presence of an insufficient partial removable denture or implant-overdenture in the opposing arch, which cannot be rendered sufficient by a reline
  * heavy smoking habit with > 20 cig/d
  * reported severe bruxism or clenching habits
  * clinically present oro-facial pain
  * depression with a Geriatric Depression Scale above 12
  * xerostomia with a stimulated salivary flow rate inferior to 0.7 ml/min
* ridge morphology type IV (Cawood and Howell, 1988)
* defects requiring bone augmentation procedures, or unhealthy soft tissues.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implant placement | 6 weeks
  Assessment of the accuracy of the methods will be based on the measure of the difference between the actual and the planned position of the mini implants, based on the measurement of (1) the global deviations at the coronal and apical regions of the mini implants, (2) the vertical deviation, and (3) the apical angle deviation. The global deviation is defined as the 3D distance between the coronal/apical centers of the planned and placed implants. The vertical deviation is the distance between the coronal center of the longitudinal axis of the planned implant and a plane parallel through the coronal center of the placed implant. The angle deviation will be measured as the angular divergence between the longitudinal axes of the planned and actual position of the mini implants. The divergence of the implant axis (in degrees) will also be recorded.
Surgery intercurrencies and complications | 6 weeks
  Any complications associated with the surgical procedures, or deviations from the prescribed protocol due to surgical intercurrences will be recorded. These include failed drilling of the planned implant site, need to raise a flap for adequate positioning of the needle drill, fracture of the bone walls, insufficient insertion torque (< 10 Ncm), early implant failure, and others.
Treatment intercurrencies and complications | Through study completion, an average of 1 year
  Any post-treatment complications associated with the use of the maxillary overdenture
Oral health-related quality of life impacts | 6 months
  Overall impacts of treatment on oral health-related quality of life will be assessed using the Oral Health Impact Profile instrument for edentulous subjects (OHIP-EDENT). It contains 19 questions in seven domains and proved to be sensitive to changes in prosthetic treatment and oral health. For each of the questions, subjects are asked how frequently they have experienced the event during the last month. Responses are given on a 5-item Likert scale. In this study, the validated Portuguese translation of the questionnaire will be utilized.
Oral health-related quality of life impacts | 1 year
  Overall impacts of treatment on oral health-related quality of life will be assessed using the Oral Health Impact Profile instrument for edentulous subjects (OHIP-EDENT). It contains 19 questions in seven domains and proved to be sensitive to changes in prosthetic treatment and oral health. For each of the questions, subjects are asked how frequently they have experienced the event during the last month. Responses are given on a 5-item Likert scale. In this study, the validated Portuguese translation of the questionnaire will be utilized.
Denture Satisfaction Index | 6 months
  Denture satisfaction will be evaluated by using the Denture Satisfaction Index (DSI; (25)), a 10mm visual analogue scale (VAS)-based questionnaire. This index evaluates ease of cleaning, general satisfaction, speech, comfort, aesthetics, stability, chewing ability, function and the general oral condition.
Denture Satisfaction Index | 1 year
  Denture satisfaction will be evaluated by using the Denture Satisfaction Index (DSI; (25)), a 10mm visual analogue scale (VAS)-based questionnaire. This index evaluates ease of cleaning, general satisfaction, speech, comfort, aesthetics, stability, chewing ability, function and the general oral condition.
Implant Survival and Success | Through study completion, an average of 1 year
  Implant Survival and Success rate will be defined as followed:
  I - Success (optimum health) II - Satisfactory survival III - Compromised survival IV - Failure (clinical absolute failure) Any of following Additionally, fractured implants will be considered as failures, except fracture of the implant apex during implant placement. Any dental implant showing excessive bone loss, such as radiolucency or infection, shall be treated in the manner best suited to the well-being of the subject, including treatment to save the dental implant.
Prosthetic Success and Survival | Through study completion, an average of 1 year
  One of the following:
  * Patrix fracture
  * Dislodged, worn or loose matrix housing
  * Matrix replacement
  * Matrix fracture
  * Fracture of the implant-supported overdenture
  * Fracture of the acrylic above a patrix
  * Fracture of denture teeth
  * Relining of implant overdenture A failure will be defined as an event leading to the loss of the reconstruction and need for the fabrication of a new overdenture.

SECONDARY OUTCOMES:
Chewing efficiency | 1-year
  Chewing efficiency will be evaluated with a two-color mixing ability test (28), where participants are given a two-colored chewing gum and are asked to chew the specimen for 20 chewing cycles. The resulting bolus is evaluated visually on a reference scale and opto-electronically using the Variance of Hue (VOH) (Halazonetis et al., 2013).
Maximum voluntary bite force (MBF) | 1-year
  The Gnathodynamometer DMD® (Kratos Equipamentos Industriais Ltda., Cotia - SP, Brazil) is utilized. It is a digital force gauge with an 8.6mm thick bite element. MBF is assessed bilaterally between the upper and lower first molar. The participant's task is to bite as hard as possible on the force gauge, but to stop clenching when she/ he starts feeling uncomfortable. A contra-lateral stabilizing element with identical thickness is used to preclude denture dislodgement. The peak force of three recordings carried out on each side will be used for analysis.
Plaque index | 1-year
  Measured at 4 sites per implant (mesial/distal/buccal/oral), according to the modified Mombelli's Plaque Index (Mombelli et al., 1987)
Bleeding on probing | 1-year
  Measured at 4 sites per implant (mesial/distal/buccal/oral), the following clinical parameters will be evaluated at baseline and each follow-up visit. Dichotomous score: yes x no
Pocket probing depth | 1-year
  Will be measured from the peri-implant mucosal margin to the bottom of the sulcus or pocket
Width of the keratinized tissue | 1-year
  The width of the keratinized tissue around implants will be measured and expressed in mm at the buccal sideated through a simple rule of three with NIH Image J V1.44.
Peri-implant bone loss | 1-year
  Intra-oral radiographs are exported and 4 parallel lines are drawn corresponding to the shoulder and the apical end of the implant on Adobe Photoshop Elements 2.0 (Adobe Systems Inc., San Jose, CA, USA). One line each is placed at the shoulder and apical end of the implant and the other two at the defined bone level on the mesial and distal aspect of the implant. Knowing the implant length and using the implant-shoulder as a reference point, bone levels can be calculated through a simple rule of three with NIH Image J V1.44.
Implant Stability - Final insertion torque | 1-year
  : after the implant is installed in its final position, the final torque of insertion will be recorded (Newtons per centimeter), as displayed during insertion with the handpiece, or measured using the manual calibrated torque gauge ratchet.
  * Peak insertion torque: maximum achieved torque value during the implant insertion (in Newtons per centimeter).
  * Periotest value: values will be categorized using the Periotest value ranges: 8 to 0: Good osseointegration; the implant can be loaded; 01 to 09: clinical examination is required; loading of the implant might or might not be possible, depending on implant type and clinical situation; 10 to 50: osseointegration is insufficient, the implant cannot be loaded.
Implant Stability - Final insertion torque | During surgery
  After the implant is installed in its final position, the final torque of insertion will be recorded (Newtons per centimeter), as displayed during insertion with the handpiece, or measured using the manual calibrated torque gauge ratchet.
Implant Stability - Peak insertion torque | During surgery
  The maximum achieved torque value during the implant insertion (in Newtons per centimeter).
Implant Stability - Periotest value | During surgery
  the Periotest® hand piece (Periotest®, Siemens AG, Bensheim, Germany) will be used with the head of the patient stabilized so that the implants were perpendicular to the floor, and the Periotest will be held parallel to the floor. The test point will be in the most gingival region of the Optiloc attachment, and each measurement will be performed 3 times and the average value will be recorded for each implant. In addition, values will be categorized using the Periotest value ranges:
  * -8 to 0: Good osseointegration; the implant can be loaded;
  * 01 to 09: clinical examination is required; loading of the implant might or might not be possible, depending on implant type and clinical situation;
  * 10 to 50: osseointegration is insufficient, the implant cannot be loaded.
Implant Stability - Periotest value | 1 year
  the Periotest® hand piece (Periotest®, Siemens AG, Bensheim, Germany) will be used with the head of the patient stabilized so that the implants were perpendicular to the floor, and the Periotest will be held parallel to the floor. The test point will be in the most gingival region of the Optiloc attachment, and each measurement will be performed 3 times and the average value will be recorded for each implant. In addition, values will be categorized using the Periotest value ranges:
  * -8 to 0: Good osseointegration; the implant can be loaded;
  * 01 to 09: clinical examination is required; loading of the implant might or might not be possible, depending on implant type and clinical situation;
  * 10 to 50: osseointegration is insufficient, the implant cannot be loaded.

CONTACTS AND LOCATIONS:
Overall Officials: Cláudio R Leles, PhD, Principal Investigator — Universidade Federal de Goias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leles CR, de Paula MS, Curado TFF, Silva JR, Leles JLR, McKenna G, Schimmel M. Flapped versus flapless surgery and delayed versus immediate loading for a four mini implant mandibular overdenture: A RCT on post-surgical symptoms and short-term clinical outcomes. Clin Oral Implants Res. 2022 Sep;33(9):953-964. doi: 10.1111/clr.13974. Epub 2022 Jul 26. PMID 35818640
- [Result] Lemos CA, Verri FR, Batista VE, Junior JF, Mello CC, Pellizzer EP. Complete overdentures retained by mini implants: A systematic review. J Dent. 2017 Feb;57:4-13. doi: 10.1016/j.jdent.2016.11.009. Epub 2016 Nov 22. PMID 27888049
- [Result] Curado TFF, Silva JR, Nascimento LN, Leles JLR, McKenna G, Schimmel M, Leles CR. Implant survival/success and peri-implant outcomes of titanium-zirconium mini implants for mandibular overdentures: Results from a 1-year randomized clinical trial. Clin Oral Implants Res. 2023 Aug;34(8):769-782. doi: 10.1111/clr.14102. Epub 2023 May 31. PMID 37254798
- [Result] Mishra SK, Chowdhary R. Patient's oral health-related quality of life and satisfaction with implant supported overdentures -a systematic review. J Oral Biol Craniofac Res. 2019 Oct-Dec;9(4):340-346. doi: 10.1016/j.jobcr.2019.07.004. Epub 2019 Aug 17. PMID 31508300
- [Result] Muller F, Duvernay E, Loup A, Vazquez L, Herrmann FR, Schimmel M. Implant-supported mandibular overdentures in very old adults: a randomized controlled trial. J Dent Res. 2013 Dec;92(12 Suppl):154S-60S. doi: 10.1177/0022034513509630. Epub 2013 Oct 24. PMID 24158342
- [Result] Feine JS, Carlsson GE, Awad MA, Chehade A, Duncan WJ, Gizani S, Head T, Lund JP, MacEntee M, Mericske-Stern R, Mojon P, Morais J, Naert I, Payne AG, Penrod J, Stoker GT, Tawse-Smith A, Taylor TD, Thomason JM, Thomson WM, Wismeijer D. The McGill consensus statement on overdentures. Mandibular two-implant overdentures as first choice standard of care for edentulous patients. Montreal, Quebec, May 24-25, 2002. Int J Oral Maxillofac Implants. 2002 Jul-Aug;17(4):601-2. No abstract available. PMID 12182304
- [Result] Thomason JM, Feine J, Exley C, Moynihan P, Muller F, Naert I, Ellis JS, Barclay C, Butterworth C, Scott B, Lynch C, Stewardson D, Smith P, Welfare R, Hyde P, McAndrew R, Fenlon M, Barclay S, Barker D. Mandibular two implant-supported overdentures as the first choice standard of care for edentulous patients--the York Consensus Statement. Br Dent J. 2009 Aug 22;207(4):185-6. doi: 10.1038/sj.bdj.2009.728. PMID 19696851
- [Result] Maniewicz S, Duvernay E, Srinivasan M, Perneger T, Schimmel M, Muller F. Effect of implant-supported mandibular overdentures versus reline on masticatory performance and salivary flow rates in very old adults-A randomized clinical trial. Clin Oral Implants Res. 2019 Jan;30(1):59-67. doi: 10.1111/clr.13392. Epub 2018 Dec 30. PMID 30500094
- [Result] Khalid T, Yunus N, Ibrahim N, Saleh NBM, Goode D, Masood M. Assessment of masticatory function of mandibular implant-supported overdenture wearers: A 3-year prospective study. J Prosthet Dent. 2020 Dec;124(6):674-681. doi: 10.1016/j.prosdent.2019.08.005. Epub 2020 Jan 15. PMID 31952858
- [Result] Boven GC, Raghoebar GM, Vissink A, Meijer HJ. Improving masticatory performance, bite force, nutritional state and patient's satisfaction with implant overdentures: a systematic review of the literature. J Oral Rehabil. 2015 Mar;42(3):220-33. doi: 10.1111/joor.12241. Epub 2014 Oct 13. PMID 25307515
- [Result] van Kampen FM, van der Bilt A, Cune MS, Fontijn-Tekamp FA, Bosman F. Masticatory function with implant-supported overdentures. J Dent Res. 2004 Sep;83(9):708-11. doi: 10.1177/154405910408300910. PMID 15329377
- [Result] Di Francesco F, De Marco G, Gironi Carnevale UA, Lanza M, Lanza A. The number of implants required to support a maxillary overdenture: a systematic review and meta-analysis. J Prosthodont Res. 2019 Jan;63(1):15-24. doi: 10.1016/j.jpor.2018.08.006. Epub 2018 Sep 28. PMID 30269880
- [Result] Di Francesco F, De Marco G, Capcha EB, Lanza A, Cristache CM, Vernal R, Cafferata EA. Patient satisfaction and survival of maxillary overdentures supported by four or six splinted implants: a systematic review with meta-analysis. BMC Oral Health. 2021 May 8;21(1):247. doi: 10.1186/s12903-021-01572-6. PMID 33962612
- [Result] Boven GC, Speksnijder CM, Meijer HJA, Vissink A, Raghoebar GM. Masticatory ability improves after maxillary implant overdenture treatment: A randomized controlled trial with 1-year follow-up. Clin Implant Dent Relat Res. 2019 Apr;21(2):369-376. doi: 10.1111/cid.12721. Epub 2019 Feb 11. PMID 30741469
- [Result] Enkling N, Saftig M, Worni A, Mericske-Stern R, Schimmel M. Chewing efficiency, bite force and oral health-related quality of life with narrow diameter implants - a prospective clinical study: results after one year. Clin Oral Implants Res. 2017 Apr;28(4):476-482. doi: 10.1111/clr.12822. Epub 2016 Mar 24. PMID 27009835
- [Result] Esposito M, Grusovin MG, Willings M, Coulthard P, Worthington HV. The effectiveness of immediate, early, and conventional loading of dental implants: a Cochrane systematic review of randomized controlled clinical trials. Int J Oral Maxillofac Implants. 2007 Nov-Dec;22(6):893-904. PMID 18271370
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Result] Allen F, McMillan A. Food selection and perceptions of chewing ability following provision of implant and conventional prostheses in complete denture wearers. Clin Oral Implants Res. 2002 Jun;13(3):320-6. doi: 10.1034/j.1600-0501.2002.130313.x. PMID 12010164
- [Result] Awad MA, Lund JP, Shapiro SH, Locker D, Klemetti E, Chehade A, Savard A, Feine JS. Oral health status and treatment satisfaction with mandibular implant overdentures and conventional dentures: a randomized clinical trial in a senior population. Int J Prosthodont. 2003 Jul-Aug;16(4):390-6. PMID 12956494
- [Result] Heydecke G, Locker D, Awad MA, Lund JP, Feine JS. Oral and general health-related quality of life with conventional and implant dentures. Community Dent Oral Epidemiol. 2003 Jun;31(3):161-8. doi: 10.1034/j.1600-0528.2003.00029.x. PMID 12752541
- [Result] Souza RF, Patrocinio L, Pero AC, Marra J, Compagnoni MA. Reliability and validation of a Brazilian version of the Oral Health Impact Profile for assessing edentulous subjects. J Oral Rehabil. 2007 Nov;34(11):821-6. doi: 10.1111/j.1365-2842.2007.01749.x. PMID 17919248
- [Result] Awad MA, Feine JS. Measuring patient satisfaction with mandibular prostheses. Community Dent Oral Epidemiol. 1998 Dec;26(6):400-5. doi: 10.1111/j.1600-0528.1998.tb01978.x. PMID 9870539
- [Result] Schimmel M, Christou P, Herrmann F, Muller F. A two-colour chewing gum test for masticatory efficiency: development of different assessment methods. J Oral Rehabil. 2007 Sep;34(9):671-8. doi: 10.1111/j.1365-2842.2007.01773.x. PMID 17716266
- [Result] Halazonetis DJ, Schimmel M, Antonarakis GS, Christou P. Novel software for quantitative evaluation and graphical representation of masticatory efficiency. J Oral Rehabil. 2013 May;40(5):329-35. doi: 10.1111/joor.12043. Epub 2013 Mar 4. PMID 23452188
- [Result] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Result] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Result] Bragger U. Use of radiographs in evaluating success, stability and failure in implant dentistry. Periodontol 2000. 1998 Jun;17:77-88. doi: 10.1111/j.1600-0757.1998.tb00125.x. No abstract available. PMID 10337315
- [Result] Bragger U, Gerber C, Joss A, Haenni S, Meier A, Hashorva E, Lang NP. Patterns of tissue remodeling after placement of ITI dental implants using an osteotome technique: a longitudinal radiographic case cohort study. Clin Oral Implants Res. 2004 Apr;15(2):158-66. doi: 10.1111/j.1600-0501.2004.00988.x. PMID 15008927
- [Result] Monje A, Ravida A, Wang HL, Helms JA, Brunski JB. Relationship Between Primary/Mechanical and Secondary/Biological Implant Stability. Int J Oral Maxillofac Implants. 2019 Suppl;34:s7-s23. doi: 10.11607/jomi.19suppl.g1. PMID 31116830